CLINICAL TRIAL: NCT05303740
Title: Efficacy and Safety of Anlotinib in the First-line or Second-line Treatment of Locally Advanced or Metastatic Esophageal Cancer in China, a Retrospective, Multicenter, Real-world Study
Brief Title: Anlotinib Retrospective Study for Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Feng Wang (Other)
Responsible Party: Sponsor-Investigator, Feng Wang, Chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: L2021-Y348-001
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — anlotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anlotinib
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — This is an observational study.

SUMMARY:
The efficacy of anlotinib in the treatment of esophageal cancer has been confirmed. The purpose of this study was to retrospectively observe the efficacy and safety of anlotinib in the first and second line of advanced esophageal cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal cancer diagnosed pathologically or clinically
* Patients who use anlotinib alone, or combined with chemoradiotherapy, or plus PD-1 inhibitors in first-line or second-line treatment

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Esophageal cancer patients previously treated with anlotinib
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
PFS | From date of admission until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
OS | From date of admission until the date of death from any cause, assessed up to 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No